CLINICAL TRIAL: NCT05833659
Title: The Comparison Between Prepectoral Breast Reconstruction and Subpectoral Breast Reconstruction Following Single-port Insufflation Endoscopic Nipple-sparing Mastectomy
Brief Title: Comparison Between Prepectoral and Subpectoral Breast Reconstruction
Acronym: RESPECT
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Health Promotion Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: RESPECT
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stage II Breast Cancer; Stage I Breast Cancer
Keywords: breast cancer; endoscopic nipple-sparing mastectomy; breast reconstruction; breast satisfaction; BREAST-Q score
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The prepectoral breast reconstruction: The patients received prepectoral breast reconstruction after single-port insufflation endoscopic nipple-sparing mastectomy
  Interventions: Procedure: The breast reconstruction method after single-port insufflation endoscopic nipple-sparing mastectomy
- The subpectoral breast reconstruction: The patients received subpectoral breast reconstruction after single-port insufflation endoscopic nipple-sparing mastectomy
  Interventions: Procedure: The breast reconstruction method after single-port insufflation endoscopic nipple-sparing mastectomy

INTERVENTIONS:
Procedure: The breast reconstruction method after single-port insufflation endoscopic nipple-sparing mastectomy — Group A:The prepectoral breast reconstruction. Group B:The subpectoral breast reconstruction

SUMMARY:
There are controversies about breast implant-based reconstruction techniques. Our center pioneered single-port insufflation endoscopic nipple-sparing mastectomy (SIE-NSM) combined with stage I prosthesis reconstruction. The study's primary objective is to compare single-port endoscopic NSM combined with pre-pectoral breast reconstruction to the subpectoral breast reconstruction group regarding breast satisfaction.

This study is an ambispective cohort study. The study will be conducted at Beijing Friendship Hospital, affiliated with Capital Medical University. Patients will be enrolled retrospectively from January 2014 to March 2022 by reviewing the medical records and recruited prospectively from March 2022 to March 2025. The two cohorts are the pre-pectoral breast reconstruction cohort and the subpectoral breast reconstruction cohort, both following single-port insufflation endoscopic nipple-sparing mastectomy. The primary outcome of this study is postoperative breast satisfaction, which the BREAST-Q score will measure. The different variables will be compared using the Χ2 test for categorical variables and the Mann-Whitney test for continuous variables.

DETAILED DESCRIPTION:
Sample size and statistical analysis This study is an ambispective cohort study. According to the previous retrospective research data of the center, the breast satisfaction score is the main research object. The standard deviation was 2.6, the non-inferiority margin was 0.15, the test level was α=0.05, β=0.2, and a one-sided test was performed. Eighty patients will be needed for two cohorts in a 1:1 ratio. Considering the 10% loss to follow-up rate, 44 patients will be required to be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with preoperative pathologically confirmed early-stage invasive breast cancer (stage I or stage II) by core needle biopsy.
2. Breast-conserving surgery is not possible due to the presence of contraindications to breast-conserving surgery, or the patient actively requests total mastectomy.
3. Patients having willingness for breast reconstruction.
4. Age between 18 to 70 years.
5. Maximum diameter of the cancer lesion ≤ 3 cm.
6. Physical examination and breast magnetic resonance imaging (MRI) confirmed that the tumor did not invade the skin, subcutaneous tissue, or chest wall.
7. The distance between the lesion and the nipple is ≥2 cm, and it is confirmed by physical examination and MRI that the nipple-areola complex is not invaded.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale of 0 to 2.

Exclusion Criteria:

1. patients having serious medical diseases, including unstable angina pectoris, myocardial infarction, and cerebrovascular accident within 6 months.
2. Having history of malignant tumor (s) within 5 years.
3. Patients under immunosuppressive therapy for organ transplantation.
4. Having continuous systemic steroid hormone therapy.
5. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with preoperative pathologically confirmed early-stage invasive breast cancer (stage I or stage II) and having willingness for breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
breast satisfaction | 12 months after operation
  measured by BREAST-Q score

SECONDARY OUTCOMES:
Physical well-being of chest | 12 months after operation
  measured by BREAST-Q score
Animation deformity | 12 months after operation
  confirmed by the doctor's physical examination
Adverse events | within 30 days after surgery
  according to Clavien-Dindo system
Local recurrence and distant metastasis of breast cancer | 12 months after operation
  physical examination or imaging examination with histologically confirmed

CONTACTS AND LOCATIONS:
Overall Officials: guoxuan gao, MD, Principal Investigator — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University
Locations (1):
- Beijing Friendship Hospital, Capital medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided